CLINICAL TRIAL: NCT04709978
Title: Redefining Community Acquired Pneumonia in Older Adults: The Role and Impact of Aspiration
Brief Title: Community Acquired Pneumonia in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Gordon and Betty Moore Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1121; Protocol Version 11/3/22 (Other: UW Madison); A534100 (Other: UW Madison); SMPH/EMERG MED (Other: UW Madison); A534255 (Other: UW Madison)
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pneumonia; Aspiration Pneumonia
MeSH Terms: conditions — Pneumonia; Pneumonia, Aspiration | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva and mouth swabs, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pneumonia: Participants will be over the age of 60 and diagnosed with pneumonia in the UW Emergency Department or treated for pneumonia in the past 6 months.
  Interventions: Diagnostic Test: Videofluoroscopic Swallowing Study; Diagnostic Test: Nuclear medicine pulmonary aspiration study; Diagnostic Test: TOR-BSST and 3 oz Water Swallow; Diagnostic Test: Sputum Culture; Diagnostic Test: MeMed BV®; Diagnostic Test: Lung Ultrasound; Diagnostic Test: Respiratory Function Tests

INTERVENTIONS:
Diagnostic Test: Videofluoroscopic Swallowing Study — Participants enrolled in supplemental study will swallow different barium containing liquid and food boluses types that are captured on fluoroscopic imaging in real time.
Diagnostic Test: Nuclear medicine pulmonary aspiration study — Participants enrolled in supplemental study will be administered radiotracer (Tc-99m-Sulfur Colloid) orally and static images of the chest will then be obtained at specified intervals over the next 2 hours to determine location of the radiotracer.
Diagnostic Test: TOR-BSST and 3 oz Water Swallow — The research specialist will conduct ten 1 tsp water swallows, one cup sip of water and a 3 ounce water swallow test with the patient. After each swallow, the participant is asked to say "ah" so that their voice quality can be assessed.
  Other Names: bedside dysphagia screening; 3 ounce water swallow test
Diagnostic Test: Sputum Culture — Patients will have sputum collected during stay (ED participants only)
Diagnostic Test: MeMed BV® — A blood test to help determine if the infection is viral or bacterial (ED participants only)
Diagnostic Test: Lung Ultrasound — To image the lungs (ED participants only)
Diagnostic Test: Respiratory Function Tests — To measure respiratory pressures.
  Other Names: manometer; peak cough flow

SUMMARY:
This study will utilize diagnostic imaging and salivary biomarkers to estimate the prevalence of aspiration in older adults with suspected community-acquired bacterial pneumonia (CABP). 150 participants over the age of 60 diagnosed with pneumonia will be recruited into this study. 62 of these participants will be enrolled in a supplemental study.

DETAILED DESCRIPTION:
Pneumonia is the most common infectious cause of mortality in older adults. Standard practice for older adults with pneumonia involves hospitalization and antibiotics. However, recent studies suggest that a significant portion of suspected community-acquired bacterial pneumonia (CABP) cases may actually be due to distinct, dysphagia-related aspiration syndromes (e.g. aspiration pneumonia, pneumonitis).

The main study will will assess whether salivary biomarkers (viscoelasticity, substance P) and swallowing function tests can be used to help differentiate CABP from aspiration-related syndromes. The following aims will be completed:

* Aim 1: Compare salivary properties and health outcomes among older adults with aspiration related pneumonia mimics and those with infectious pneumonia
* Aim 2: Compare appearance of lung ultrasound findings among older adults with aspiration related pneumonia mimics and those with infectious pneumonia.
* Aim 3: Describe dysphagia screening results, patient reported swallowing function, salivary properties, oral/nasopharyngeal microbiome profiles, in older adults with pneumonia presenting to the ED.
* Aim 4: Assess the potential impact of the MeMed BV® test's result on patient management decision making, including antibiotic prescribing and disposition.

A supplemental study will be the first to utilize diagnostic imaging (videofluoroscopic evaluation of swallowing and radionuclide salivagram) to estimate the prevalence of aspiration in older adults with suspected CABP.

* Aim 1: Determine the prevalence of dysphagia-related aspiration among older adults with pneumonia.

ELIGIBILITY:
Emergency Department (ED) Recruitment

Inclusion Criteria:

* 60 years of age or older
* Patient has clinical criteria for pneumonia or is being treated for pneumonia as defined by abnormal chest imaging or receiving antibiotics for a chest infection or the provider thinks the patient has pneumonia or is planning to treat the patient for pneumonia.
* Patient is clinically stable and able to safely drink water, per the emergency department provider
* Ability to provide consent or the presence of a legally authorized representative (LAR) who can consent on behalf of the patient

Exclusion Criteria:

* Prisoner
* Non-English speaking
* Respiratory symptoms for 7 days or more

Phone Recruitment

Inclusion Criteria:

* 60 years of age and older
* Patient was diagnosed with or treated for pneumonia at UW Health in the past 6 months
* Ability to provide consent or the presence of a legally authorized representative (LAR) who can consent on behalf of the patient

Exclusion Criteria:

* Prisoner
* Non-English speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from the UW Emergency Department and via phone, 60 years of age or older diagnosed with or treated for pneumonia in the past 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Aspiration | up to 6 months on study
  As defined by VFSS and radionuclide salivagram imaging studies.

SECONDARY OUTCOMES:
Salivary extensional viscosity | Any point during follow up within 6 months of index visit
  Extensional viscosity will be determined using an extensional rheometer (Thermo-Fisher CaBER) and will be recorded 3 times per sample.
Salivary Substance P Concentration | Any point during follow up within 6 months of index visit
  Substance P is a salivary protein
Salivary pH | Any point during follow up within 6 months of index visit
  Salivary pH will be measured using a digital pH meter.
Recurrent pneumonia | Any point during follow up within 6 months of index visit
  As assessed on medical chart review
Lung Ultrasound Findings for ED participants | at ED visit, baseline
  Lung ultrasound exams will be compared between older adults with aspiration related pneumonia mimics and those with infectious pneumonia. Interpretation of ultrasound images will be performed by two ultrasound fellowship trained EM faculty, blinded to any clinical information. Each lung ultrasound view captured will be reviewed and interpreted descriptively. Lung ultrasound findings will be described with the following features: crisp or irregular pleural line, A line artifacts, isolated Z line artifacts, static air bronchograms, dynamic air bronchograms, tissue-like consolidation without bronchograms, coalescent B lines (presence and how many per interspace), discrete B lines (presence and how many per interspace), subpleural hypoechoic consolidation, and pleural effusion.
Patient Reported Swallowing Function as measured by physical symptoms on SWAL-QOL | at Point of Care visit, up to 6 months
  All participants will complete self report surveys at their first study visit. The physical symptoms question on the SWAL-QOL asks the participant to identify how often they experienced specific symptoms in the past month, from 1 (almost always) to 5 (never). The total score is transposed to 0-100 with higher scores indicating better swallowing function.
Percent Viral vs. Bacterial Infection for ED participants | at ED visit, baseline
  MeMed BV® test results for participants recruited in the ED.
Respiratory Pressure | Any point during follow up within 6 months of index visit
  Maximum expiratory pressure and maximum inspiratory pressure will be measured using a handheld digital manometer. This test will take approximately 5 minutes.
Peak Expiratory Flow (PEF) | Any point during follow up within 6 months of index visit
  A handheld digital peak cough flow meter will be used to assess PEF to quantify cough function. This test will take approximately 3 minutes.
Forced Expiratory Volume (FEV1) | Any point during follow up within 6 months of index visit
  A handheld digital peak cough flow meter will be used to assess forced expiratory volume (FEV1) to quantify cough function. This test will take approximately 3 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pulia, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No